CLINICAL TRIAL: NCT00791180
Title: Clinical Outcomes Following Posterior Lateral Fusion With the Dynesys(R) Spinal System
Brief Title: Posterior Lateral Fusion (PLF) With Dynesys
Status: Completed | Type: Observational
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Other Study IDs: 2006-002
Record Dates: First submitted 2008-11-13; First posted 2008-11-14 (Estimated); Last update posted 2011-09-29 (Estimated); Status verified 2011-09

CONDITIONS: Spondylolisthesis
Keywords: dynamic stabilization; Dynesys; fusion success; Immobilization of spinal segments as an adjunct to fusion in the treatment of the following:; acute and chronic instabilities or deformities of the thoracic, lumbar, and sacral spine; degenerative spondylolisthesis with objective evidence of neurologic impairment; failed previous fusion (pseudarthrosis).
MeSH Terms: conditions — Spondylolisthesis; Pseudarthrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The primary purpose of this study is to track and document the clinical outcomes of patients with radicular pathology following posterior lateral fusion with the Dynesys Spinal System. Secondary purpose of this study is to assess outcomes with historical controls along a continuum of motion and anatomy sparing procedures.

DETAILED DESCRIPTION:
This study will help the patient to the extent that it will allow the comparison of this unique treatment to the corpus of literature on radicular pathology, thus focusing a specific treatment for a specific pathology.

ELIGIBILITY:
Inclusion Criteria:

* Spondylolisthesis of less than Grade II at the index level (degenerative with intact pars)
* Will receive a decompression for lumbar stenosis
* Symptoms of leg and/or back pain
* One pathological level
* Between the ages of 20 and 80 at the time of surgery
* Non-responsive to non-surgical treatment for at least six months

Exclusion Criteria:

* Osteolytic spondylolisthesis
* Planned complete facetectomy
* Two or more pathological levels (and as enumerated int he Dynesys Spinal system instructions for use)
* Use in the cervical spine
* Active systemic or local infection
* Extreme obesity as defined by a Body Mass Index (BMI)over 40. BMI calculated using Appendix A, adapted from the National Heart, Lung, and Blood Institute, Clinical Guidelines on the Identification, Evaluation, and Treatment of Overweight and Obesity in Adults.
* Pregnancy
* Mental illness
* Severe osteoporosis or osteopenia. The World Health Organization defines osteoporosis as BMD<-2.5t. Professional discretion should be used and if bone quality is in question a DEXA scan is recommended.
* Sensitivities/allergy to metals, polymers, polyethylene, polycarbonate urethane and polyethylene terephthalate
* Alcohol or drug abuse
* Patient unwilling or unable to follow postoperative instructions
* Soft tissue deficit not allowing sound closure
* Any medical or physical condition that would preclude the potential benefit of spinal surgery
* Inadequate pedicles of the lumbar or sacral vertebrae; congenital abnormalities, tumors or other conditions that would prevent secure component fixation that has the potential to decrease the useful life of othe devices;
* Any medical or mental condition which would exclude the patient at high risk from surgery of the severity

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Clinical outcomes following postierior lateral fusion with the Dynesys(R) Spinal System
Sampling Method: Non-Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2006-03; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Clinical Outcomes | Pre-op, Surgery, 3 month, 6 month, 12 months and 24 months

SECONDARY OUTCOMES:
Surgical Outcomes | Pre-op, Surgery, 3 months, 6 months, 12 months and 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Jozef Murar, M.D., Study Director — Zimmer Spine
Locations (1):
- Foundation Surgical Hospital, Houston, Texas, United States